CLINICAL TRIAL: NCT03670537
Title: Iron Parameters in Non-anemic First Trimester Gravidas
Status: Completed | Type: Observational
Sponsor: Auerbach Hematology Oncology Associates P C (Other)
Collaborators: MedStar Women's Care at Honeygo (Unknown)
Responsible Party: Principal Investigator, Michael Auerbach MD, President and Clinical Professor of Medicine, Georgetown, Auerbach Hematology Oncology Associates P C
Other Study IDs: Protocol 3
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Results first posted 2018-10-15 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Iron Deficiency (Without Anemia); Pregnancy
Keywords: Iron deficiency, Non-anemic; Pregnancy
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First trimester pregnant women
  Interventions: Diagnostic Test: Iron parameters

INTERVENTIONS:
Diagnostic Test: Iron parameters — Serum iron, total iron binding capacity, TSAT (Fe/TIBC), serum ferritin

SUMMARY:
The purpose of the study is to see the percentage of non-anemic, first trimester gravidas presenting to their obstetricians, who are iron deficient.

DETAILED DESCRIPTION:
The 2015 United States Preventive Services Task Force (USPSTF) stated "there is insufficient evidence to recommend the routine screening for iron deficiency in non-anemic gravidas". The basis for this recommendation is the lack maternal or fetal outcome data in this population. To date, there are no guidelines for the treatment of non-anemic, iron deficiency pregnancy women with or without anemia. Obstetricians and gynecologists often do not screen for iron deficiency unless the mean corpuscular volume (MCV) is reduced even in the presence of a reduced hemoglobin. Iron deficiency occurs prior to a decrement in hemoglobin concentration, followed by a decrease in the MCV which occurs after. Subsequently, if these recommendation are followed up to 50% of iron deficient pregnant women remain undiagnosed.

While prospective studies may be absent proving that routine screening and supplementation is beneficial, there is ample evidence that iron deficiency in mothers and infants results in significant morbidity, even in the absence of anemia. Fetal, neonatal and childhood brain growth and development require iron, with deficiencies resulting with adverse effects on myelination, neurotransmitter synthesis and brain programming. There is a two-fold incidence of preterm birth, three-fold increase in low birth weight and small for gestational age infants. In addition to negative effects on the fetus, maternal iron deficiency is associated with an increased risk for caesarean delivery, transfusion, perinatal bleeding, pre-eclampsia, placental abruption, poor wound healing, cardiac failure and even death. Of note, using existing guidelines infants are not screened for iron deficiency even if they are at high risk (preterm, infants of diabetic mothers, smokers or those with intrauterine growth restriction.

Published evidence suggests that when iron deficiency is present later in pregnancy in the mother, adequate iron delivery to the fetus does not occur. In a prospective study of 2400 urban women with iron deficiency in the second and third trimesters, while supplementation resulted in a significant improvement in maternal hemoglobin concentrations and iron parameters, over 45% of infants were iron deficient at birth.

Subsequently, while prospective studies are lacking supporting routine screening and iron supplementation, high quality published evidence imputing a litany of morbid events associated with iron deficiency, calls into question the recommendations of the USPSTF. Until such evidence is available based on the preponderance of evidence supporting absence of harm with either screening or supplementation we believe all gravidas presenting to their obstetricians should be screened for iron deficiency.

We propose a prospective observation study of one hundred consecutive, non-selected, non-anemic, first trimester pregnant women to have iron parameters added to their routine laboratory tests. While we realize this is not standard, many practices already have adopted this screening process. We intend to redact all demographic patient information and expect to incur no uncovered costs. As a result we believe neither investigational review board or informed consent is necessary. In hundreds of patients so screened we have encountered no insurance pushback. The additional tests will include only serum iron, total iron binding capacity (TIBC), percent transferrin saturation (Fe/TIBC) and serum ferritin. The data will be stratified by parity.

We anticipate to find an incidence of iron deficiency of 30-40% based on either a low TSAT or low serum ferritin. Such a finding should motivate properly powered, prospective outcome analyses supporting a new paradigm that incorporating the low cost screening for iron deficiency accompany standard screening tests at the beginning of pregnancy irrespective of the presence or absence of anemia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant in first trimester
* Non-anemic

Exclusion Criteria:

* anemia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women presenting to their obstetricians
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Auerbach Hematology and Oncology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Auerbach M, Abernathy J, Juul S, Short V, Derman R. Prevalence of iron deficiency in first trimester, nonanemic pregnant women. J Matern Fetal Neonatal Med. 2021 Mar;34(6):1002-1005. doi: 10.1080/14767058.2019.1619690. Epub 2019 Jun 3. PMID 31154873

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | First Trimester Pregnant Women
Started | 102
Completed | 101
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | First Trimester Pregnant Women
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 101
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 101
Gravidity (number of pregnancies) [Count of Participants; unit: Participants]
  Gravida 1 | 29
  Gravida 2 | 30
  Gravida 3 | 23
  Gravida 4 | 11
  Gravida 5 | 6
  Gravida 6 or more | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent of Non-anemic Patients With Iron Deficiency Stratified by Gravidity
Description: Either low serum ferritin or low percent transferrin saturation (TSAT)
Time Frame: Day 1 presentation to obstetrician
Measure: Count of Participants; unit: Participants
Arm/Group | First Trimester Pregnant Women
Number analyzed (Participants) | 101
Participants
  Serum ferritin 25-30ng/ml | 9
  Serum ferritin 20-25ng/ml | 3
  Serum ferritin <20ng/ml | 6
  TSAT <19% | 38

ADVERSE EVENTS:
Time Frame: During blood draw
Arm/Group | First Trimester Pregnant Women
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT03670537/Prot_SAP_000.pdf